CLINICAL TRIAL: NCT04364607
Title: Intramuscular Neostigmine for Accelerating Bladder Emptying After Cesarean Section by Spinal Anesthesia
Brief Title: IM Neostigmine for Accelerating Bladder Emptying After CS by Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS.19.12.937.R1
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Cesarean Section Complications
Keywords: Cesarean Section; Spinal anesthesia; Postoperative urine retention (POUR)
MeSH Terms: interventions — Neostigmine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neostigmine group (Active Comparator): After cesarean delivery, women will receive 0.5 mg IM neostigmine
  Interventions: Drug: Neostigmine
- Placebo group (Placebo Comparator): After cesarean delivery, women will receive IM NaCl 0.9% as a placebo
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Neostigmine — Participants will receive 0.5 mg IM neostigmine
  Other Names: Epistigmin
  Arms: Neostigmine group
Drug: NaCl 0.9% — Participants will receive IM NaCl 0.9% as a placebo
  Other Names: Normal Saline
  Arms: Placebo group

SUMMARY:
The aim of this study is to assess the efficacy of IM neostigmine (0.5 mg) for acceleration of bladder evacuation and prevention of postoperative urine retention following cesarean delivery carried out under spinal anesthesia

DETAILED DESCRIPTION:
Following cesarean delivery, women will receive either 0.5 mg IM neostigmine (study group) or IM NaCl 0.9% (control group). Bladder ultrasonography will be done every hour until spontaneous voiding occurs. If postoperative urine retention occurred (void inability with bladder volume > 600 ml by ultrasound), urinary catheterization will be done.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing elective cesarean deliver under spinal anesthesia.

Exclusion Criteria:

* The age of the patient is more than 35 years of less than 20 years.
* The body mass index of the patient is more than 35 kg/m2 or her height is more than 180 cm or less than 150 cm.
* Multiple gestation.
* The patient is in active labor.
* Vaginal bleeding, placenta previa or abruption of the placenta.
* Presence of fetal distress.
* Urinary symptoms.
* Medical disorders co-existing with or complicating pregnancy.
* Contraindications for or history of adverse reaction of Neostigmine.
* Contraindication for spinal anesthesia.
* Refusal of the patient to receive spinal anesthesia.
* Intraoperative significant hemorrhage.
* Duration of the operation is more than one hour.
* Occurrence of postoperative complications as eclampsia.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Time to first voiding after treatment | Until 12 hours postoperatively
  Time interval between IM injection of neostigmine or NaCl and occurrence of first voiding
Time to first voiding after catheter removal | Until 12 hours postoperatively
  Time interval between catheter removal and occurrence of first voiding

CONTACTS AND LOCATIONS:
Overall Officials: Aml M Aljaml, Principal Investigator — Mansoura University; Mohamed A Elnegery, MD, Study Director — Mansoura University; Nermeen M Shams-Eldien, MD, Study Director — Mansoura University; Khalid Samir, MD, Study Director — Mansoura University; Mohamed S Abdelhafez, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication and forever
Access Criteria: Contact to corresponding author